CLINICAL TRIAL: NCT04236687
Title: Prospective, Controlled Investigation of Prostate Artery Embolization Compared to Holmium Laser Enucleation of the Prostate for the Treatment of Symptomatic Benign Prostatic Hyperplasia
Brief Title: Prostate Artery Embolization Compared to Holmium Laser Enucleation of the Prostate for Benign Prostatic Hyperplasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HBP01
Record Dates: First submitted 2020-01-15; First posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Holmium laser enucleation of the prostate (Experimental): Holmium laser will be used to enucleate the prostatic hyperplasia trough the urethra
  Interventions: Device: Holmium laser enucleation of the prostate
- Artery embolization of the prostate (Active Comparator): A catheter is placed in the prostate artery, a fluid containing thousands of tiny particles (microspheres) is injected through the catheter into these small arteries which nourish the prostate. The injected microspheres will slow the blood flow to the prostate.
  Interventions: Procedure: Artery embolization of the prostate

INTERVENTIONS:
Device: Holmium laser enucleation of the prostate — Holmium laser will be used to enucleate the prostatic hyperplasia trough the urethra
  Arms: Holmium laser enucleation of the prostate
Procedure: Artery embolization of the prostate — A catheter is placed in the prostate artery, a fluid containing thousands of tiny particles (microspheres) is injected through the catheter into these small arteries which nourish the prostate
  Arms: Artery embolization of the prostate

SUMMARY:
The purpose of this study is to evaluate improvement of symptoms from benign prostatic hyperplasia (BPH) as assessed by the International Prostate Symptom Score (IPSS) for prostate artery embolization (PAE) with microspheres (Embozene™, 400µm) compared to conventional Holmium laser enucleation of the prostate (HoLEP).

DETAILED DESCRIPTION:
This is a prospective randomized controlled study that collects data of patients with benign prostatic hyperplasia that are treated with prostatic artery embolization (PAE) or with Holmium laser enucleation of the prostate (HoLEP). For PAE a catheter is placed in the prostate artery, a fluid containing thousands of tiny particles (microspheres) is injected through the catheter into these small arteries which nourish the prostate. The injected microspheres will slow the blood flow to the prostate. For HoLEP a Holmium laser will be used to enucleate the prostatic hyperplasia trough the urethra. Clinical follow-up include clinical visit after 1, 6 and 12 months. Acute as well as long term complications will be recorded. The patients fill in the questionnaires for urologic disease. Urodynamic examination will record functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients evaluated in the urology department and candidates to surgical treatment
* Age > 45 years
* IPSS ≥ 10
* Maximum urinary flow < 12 milliliters (mL)/second (s)
* Post-void residual urinary volume < 300mL
* Prostatic volume between 20mL and 250mL assessed by ultrasound
* Signed informed consent

Exclusion Criteria:

* PSA > 10 (if not negative prostate biopsy)
* Life expectancy below 1 year
* Renal insufficiency defined as Glomerular Filtration Rate < 30 ml/min/1,73m2
* Known severe reactions to iodine-based contrast or gadolinium-based contrast
* CT examination reveals no access to the prostate arteries.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of symptoms assessed by International Prostate Symptom Score (IPSS) | Baseline to 6 months after procedure
  Change in prostatic symptoms using the International Prostate Symptom Score (IPSS). IPSS score goes from 0 to 35. Higher values mean worse outcome (prostate symptons)

SECONDARY OUTCOMES:
Maximum urinary flow | Baseline to 6 months after procedure
  Maximum urinary flow rate (Qmax). Evaluated in milliliter per seconds (mL/s).
Post-void residual urinary volume | Baseline to 6 months after procedure
  Post-void residual urinary volume (PVR). Post-void urinary volume: evaluated in milliliters (mL)
Prostate specific antigen (PSA) | Baseline to 6 months after procedure
  Determination in plasma of the prostate specific antigen (PSA)
Procedure related adverse events | Baseline to 6 months after procedure
  Evaluation of Procedure related adverse events assessed by Clavien-Dindo modified score. Clavien Dindo modified score: the score goes from 1 to 5. Higher values mean worse outcome (surgical complications)
Procedure related effects on sexual function | Baseline to 6 months after procedure
  Changes in sexual function assessed by International Index of Erectile Function (IIEF) score. IIEF: the score goes from 6 to 75. Lower values mean worse outcome (overall male sexual function).
Procedure related effects on urinary continence | Baseline to 6 months after procedure
  Changes in urinary continence assessed by the International Consultation on Continence Questionnaire Short Form (ICIQ-SF). ICIQ-SF: score goes from 0 to 21. Higher values mean worse outcome (urinary continence)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Agreda, MD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided